CLINICAL TRIAL: NCT02817932
Title: A Single-center, Open-label, Ascending Single- and Multiple-oral Dose Study to Evaluate the Pharmacokinetics and Safety of Ranolazine PR in Healthy Korean and Caucasian Male Subjects
Brief Title: A Study of Pharmacokinetics and Safety of Ranolazine PR in Healthy Korean and Caucasian Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.Menarini Asia-Pacific Holdings Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAKR/15/Ran-Ang/001
Record Dates: First submitted 2016-04-29; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Male Individuals
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Korean, 375 mg) (Experimental): Group 1 (Korean, 375 mg): Ranolazine PR 375 mg
  Interventions: Drug: Ranolazine
- Group 2 (Korean, 500 mg): (Experimental): Group 2 (Korean, 500 mg): Ranolazine PR 500 mg
  Interventions: Drug: Ranolazine
- Group 3 (Korean, 750 mg): (Experimental): Group 3 (Korean, 750 mg): Ranolazine PR 750 mg
  Interventions: Drug: Ranolazine
- Group 4 (Caucasian, 375mg) (Experimental): Group 4 (Caucasian, 375mg) : Ranolazine PR 375 mg
  Interventions: Drug: Ranolazine
- Group 5 (Caucasian, 750mg) (Experimental): Group 5 (Caucasian, 750mg) : Ranolazine PR 750 mg
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine

SUMMARY:
The purpose of this study is:

To assess the pharmacokinetic profile and safety of ranolazine PR in healthy Korean and Caucasian volunteers after oral administration of Ranolazine at the doses of 375, 500, 750mg after single and repeated oral administrations.

DETAILED DESCRIPTION:
Ranolazine is an antianginal drug that exerts its effects by inhibition of the late sodium current in cardiac cells. This action reduces intracellular sodium accumulation and consequently decreases intracellular calcium overload which is expected to reduce myocardial stiffness, oxygen consumption and ATP utilization and improve blood flow to the microvasculature.These effects of ranolazine do not depend upon reductions in heart rate or blood pressure or vasodilation.

Ranolazine PR, approved for treatment of chronic angina in 56 countries and currently marketed in 21 countries including the US shows clinical efficacy and tolerability in the proposed therapeutic dose range from 375 mg to 750mg. Factors that may affect ranolazine pharmacokinetics including demographics, drug-drug interactions, disease state, CYP2D6 metabolizer genotype status and impaired renal or hepatic functions have been studied. The relationship between ranolazine plasma concentration and clinical effects has been also well-established. This PK study has been designed as a bridging study for Ranolazine PR registration in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult Korean or Caucasian males, 19 - 45 years of age

   * Korean subjects: first generation of Korean subject born in Korea, both parents and the four grandparents must be of Korean origin. Proof of Korean ethnicity will be documented by medical interview and appropriate materials (e.g. Korean passport, Korean resident card) will be retained in the subject's folder
   * Caucasian subjects: first generation of Caucasian subject, both parents and the four grandparents of European descent. Documentation of ethnicity will be by medical interview and by appropriate materials (e.g. passport, birth certificate(if not available, a signed affirmation by the subjects)) will be retained in the subject's folder
2. Subjects weighing ≥ 50 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit
3. Subjects with no clinically significant abnormal findings as determined by physical examination, ECG, medical history, or clinical laboratory test results
4. Subjects who agreed to voluntarily participate in this study and comply with all the study requirements by signing informed consent form after being informed of the nature of this study and understanding all aspects of this study

Exclusion Criteria:

1. History of clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorder
2. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
3. Relevant chronic or acute infections
4. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
5. Administration of any investigational products within 3 months from the first dose of the study drug (ranolazine PR)
6. History of participating other BE study or clinical trial within 3 months from the first dose of the study drug(ranolazine PR)
7. Any of the following vital sign abnormalities

   * Systolic blood pressure: <90 mmHg or >140 mmHg
   * Diastolic blood pressure: <50 mmHg or > 90 mmHg
   * Pulse rate: <50 bpm or >90 bpm
8. Any of the following ECG abnormalities

   * PR > 210 msec
   * QRS complex > 120 msec
   * QTcF > 430 msec
9. Any finding in the physical examination deviating from normal and judged clinically significant by the investigator
10. Any laboratory value outside of the reference range that the investigator considers to be of clinical significance
11. Subjects who have donated blood or received blood transfusion within 90 days of participating in this study
12. Subjects who are positive for Hepatitis B, Hepatitis C, VDRL and HIV
13. Subjects who showed positive result in alcohol and drug abuse tests
14. Subjects who have smoked over 10 cigarettes until 90 days prior to the study initiation or who is not able to stop smoking throughout the hospitalization period
15. Subjects who took prescribed medications within 14 days or over-the-counter (OTC) medications within 7 days prior to the first dose of the study drug (ranolazine PR) or who have to take these medications during the study period
16. Subject who judged not eligible for study participation by investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic assessment | Up to 5 days
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic Assessment | Up to 5 days
  Plasma concentration (maximum,through, average)
Pharmacokinetic Assessment | Up to 5 days
  Tmax
Pharmacokinetic Assessment | Up to 5 days
  Half-life

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events assessed using MedDRA | 5 days
  Assessment based on reported symptoms, physical examination, vital signs, adverse events, ECGs, laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo H, Lee SW, Yoon DY, Yoon SH, Cho JY, Yu KS, Jang IJ, Lee S. Pharmacokinetics and Safety of Extended-release Ranolazine in Korean and White Healthy Subjects. Clin Ther. 2021 Mar;43(3):526-534.e4. doi: 10.1016/j.clinthera.2021.01.005. Epub 2021 Jan 29. PMID 33518355